CLINICAL TRIAL: NCT07199790
Title: Effect of Action Observation Combined With Therapeutic Exercise on Balance and Falls in Community-Dwelling Adults ≥65: A Randomized Trial
Brief Title: Action Observation and Exercise for Balance in Older Adults: A Randomized Trial.
Acronym: AOBAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Tania López Hernández, Phd, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09/2025
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Balance Disorders; Fall; Elderly (People Aged 65 or More); Exercise; Observation; Physical Therapist
Keywords: balance; strength; referent; exercise therapy; healthy aging; action observation
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Intervention: Control Group (No Intervention): Participants will not engage in any therapeutic exercise program or action observation.
- Exercise Group (Experimental): Participants will perform a therapeutic exercise program aimed at improving balance and preventing falls, three times per week for twelve weeks.
  Interventions: Other: Therapeutic exercise
- Standard Referent Group (Experimental): Participants will perform the same therapeutic exercise program aimed at improving balance and preventing falls, three times per week for twelve weeks. In addition, they will observe a standard model performing the same program, also three times per week.
  Interventions: Other: Action observation videos; Other: Therapeutic exercise
- Self-Selected Referent Group (Experimental): Participants will perform the therapeutic exercise program aimed at improving balance and preventing falls, three times per week for twelve weeks. In addition, they will observe a model they have personally selected based on perceived similarity, also three times per week, performing the same program.
  Interventions: Other: Action observation videos; Other: Therapeutic exercise

INTERVENTIONS:
Other: Action observation videos — The participant will see videos of balance exercises performed by the assigned reference, depending on their group, without performing any physical movement.
  Arms: Self-Selected Referent Group; Standard Referent Group
Other: Therapeutic exercise — The therapeutic exercise program aimed at improving balance and preventing falls will be carried out three times per week (Monday, Wednesday, and Friday), with each session lasting 30-45 minutes. Each session will be structured into three blocks: a warm-up of 5-10 minutes, a main block focused on balance and strength lasting 20-25 minutes, and a cool-down of 5-10 minutes.
  Arms: Exercise Group; Self-Selected Referent Group; Standard Referent Group

SUMMARY:
The primary objective is to evaluate the effectiveness of combining action observation with a therapeutic exercise program to improve balance and prevent falls in adults aged ≥65 with low to moderate fall risk.

DETAILED DESCRIPTION:
Background: Action observation activates brain networks involved in motor learning and has shown benefits in neurological and musculoskeletal populations (improvement of balance, gait, and pain). However, evidence in older adults at risk of falls and the role of the observed model remain underexplored. Objectives: The primary objective is to evaluate the effectiveness of combining action observation with a therapeutic exercise program to improve balance and prevent falls in adults aged ≥65 with low to moderate fall risk. Secondary objectives include comparing efficacy according to the observed model, and analyzing effects on strength, fear of falling, adherence, and fall incidence. Methods: A single-blind, randomized clinical trial of 24 weeks (12 intervention, 12 follow-up) is planned. A total of 104 participants will be allocated to four groups: control, exercise, exercise with action observation of a standard model, and exercise with action observation of a self-selected model. The intervention (therapeutic exercise program and/or action observation of the same program) will be delivered three times per week with biweekly progressions. The primary outcome will be balance (static balance measured by sway area on force platform and dynamic balance assessed by Timed Up and Go test). Secondary outcomes will include handgrip and lower limb strength, fear of falling, adherence, and fall incidence. Assessments will be conducted at weeks 0, 4, 8, 12, and 24. Both ITT and per-protocol analyses will be performed, with intra- and inter-group comparisons (p<0.05). Discussion: If effective, this low-cost, low-technology program could be easily scaled up in primary care and community settings, with potential impact on public health and physiotherapy. Applicability may also extend to neurorehabilitation and secondary prevention in frailty. Anticipated limitations: adherence, partial blinding, and external validity limited to community-dwelling older adults. Implications: development of concise practice guidelines, standardized audiovisual materials, and future research in clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 65 years of age with low or moderate risk of falls as measured by the Timed Up and Go test, who have voluntarily signed the informed consent form and are willing to follow the protocol proposed by the research team.

Exclusion Criteria:

* Presence of uncorrected visual impairments preventing screen observation; diagnosis of a condition that makes adherence to the protocol impossible (cognitive, oncological, psychiatric, psychological, vestibular, neurological, etc.); presence of a musculoskeletal injury at the time of selection and/or prior participation in studies involving movement representation methods.

Withdrawal criteria: Lack of participant compliance, defined as failure to complete at least 80% of the intervention sessions and assessments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Static balance | 12 weeks
  Center of pressure analysis: The displacement of the center of pressure (CPD) of the participants will be measured through posturographic tests performed on a force platform. The following variables related to the center of pressure (CoP) will be calculated: the roll area (in square millimeters) and the distribution of the weight load on both sides.
Dynamic balance | 12 weeks
  To assess participants' dynamic balance, the Timed Up and Go test (39-41) will be used. This test records the time, in seconds, it takes for an individual to rise from a chair, walk three meters, turn around, return, and sit down again. It is one of the most widely used tools in older adults due to its simplicity, quick administration, and high reliability. Intra- and inter-rater reliability values range from 0.94 to 0.99, and test-retest reliability from 0.95 to 0.99. Moreover, it shows significant correlations with lower-limb strength, the Berg Balance Scale, and other functional assessments.

SECONDARY OUTCOMES:
Trunk and lower extremity muscle strength | 12 weeks
  Analogue dynamometry will be used as an evaluation method and will be recorded in Newtons (N) with the Saehan SKU SH5007 back, leg and chest dynamometer.
Satisfaction assessed by a selfcreate questionnaire | 12 weeks
  A questionnaire specifically designed to evaluate participants' satisfaction with their experience in the study will be used once they have completed their participation.
Grip strength | 12 weeks
  A digital dynamometer will be used as the assessment method, and results will be recorded in kilograms using the K-Grip hand dynamometer (K-Invent®, Montpellier, France) through the grip strength test. Three 3-second trials will be performed with each hand, with 30 seconds of rest between attempts, and the best result will be selected.
Safety and fear of falling | 12 weeks
  The validated Spanish version of the Short Falls Efficacy Scale-International (Short FES-I) will be used. This scale comprises 7 items related to daily life activities, each rated on a 4-point scale: not at all concerned (1 point), somewhat concerned (2 points), fairly concerned (3 points), or very concerned (4 points). The total score ranges from 7 to 28, with higher scores indicating greater fear of falling. The Short FES-I has shown high internal consistency (Cronbach's alpha = 0.90; intraclass correlation coefficient = 0.89), good test-retest reliability (Spearman's rho = 0.76), and strong concurrent criterion validity, as evidenced by its high correlation with the original FES-I (Spearman's rho = 0.90).
Adherence | 12 weeks
  Adherence will be evaluated by calculating the ratio between the number of sessions completed and the total number of sessions scheduled. Recording will be carried out using a weekly log sheet filled out by participants and supervised by the research team.
Incidence of falls | 12 weeks
  Fall events will be recorded through self-reporting during the entire intervention and follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultat de Medicina i Ciències de la Salut, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrose AF, Paul G, Hausdorff JM. Risk factors for falls among older adults: a review of the literature. Maturitas. 2013 May;75(1):51-61. doi: 10.1016/j.maturitas.2013.02.009. Epub 2013 Mar 22. PMID 23523272
- [Background] Zhang M, Zhang T, He Y, Luo J. Comparison of motor imagery and action observation on lower limb function in older adults: a systematic review and meta-analysis. Geriatr Nurs. 2025 Sep-Oct;65:103468. doi: 10.1016/j.gerinurse.2025.103468. Epub 2025 Jul 5. PMID 40618719
- [Background] Leem SH, Kim JH, Lee BH. Effects of Otago exercise combined with action observation training on balance and gait in the old people. J Exerc Rehabil. 2019 Dec 31;15(6):848-854. doi: 10.12965/jer.1938720.360. eCollection 2019 Dec. PMID 31938708
- [Background] Lopez Hernandez T, Caparo Ferre M, Salas-Huetos A, Salvat Salvat I, Adillon Camon C. Influence of referent selection on balance in action observation: A randomized controlled trial. Complement Ther Med. 2025 Jun;90:103150. doi: 10.1016/j.ctim.2025.103150. Epub 2025 Feb 20. PMID 39986658